CLINICAL TRIAL: NCT00599456
Title: A Placebo Controlled Double Blinded Prospective Study to Investigate the Usefulness of Omega 3 Fatty Acids in the Relief of Vasomotor Symptoms of Menopausal Women
Brief Title: Investigation of the Usefulness of Omega 3 Vitamins in the Relief of Hot Flashes in Menopausal Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27103
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Hot Flashes; Menopause
Keywords: Hot flashes; Menopause; Omega 3 fatty Acids
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Omega 3 vitamin supplements
  Interventions: Dietary Supplement: Omega 3 fatty acid vitamins
- 2 (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acid vitamins — Omega 3 fatty acid vitamins, 2 capsules, by mouth, daily, for 3 months
  Arms: 1
Dietary Supplement: Placebo capsules — Placebo capsules,2 capsules, by mouth, daily for 3 months
  Arms: 2

SUMMARY:
Hot flashes can be a disturbing symptom of menopause. Prescription medications are commonly used for symptom relief. Several non-prescription therapies are under investigation. This study will examine the use of omega-3 (fish oil) supplements to see if it helps relieve hot flashes and therefore improve the quality of life.

Study Hypotheses:

Menopausal women who take Omega 3 vitamins(fish oils)will show improvement in the severity of their hot flashes.In addition women who take Omega 3 supplements will show improvement in their lipid profiles.

DETAILED DESCRIPTION:
This study requires you to have blood drawn twice, record your hot flashes for a total of 3 weeks, and to take a product every day for 12 weeks. It will also entail 4 visits and up to 4 telephone contacts. The information you provide will be maintained in a database accessible only to the primary investigator and research team. You will be assigned a code number for your blood work and all other information. The key to this code will be maintained in this database.

Overall 60-100 women will be recruited for this study locally. During the course of the study you will get overall two blood draws amounting to up to a teaspoon for measurement of your cholesterol and fat levels.

This project consists of three phases.

Phase I

We will ask you questions about your medical history and your health. You will then be asked to provide a urine sample which will be used to confirm your menopausal status with a FSH level. You will be requested to keep a record of your hot flashes for one week using a symptom diary. Upon completion of the diary, you will return to the study site. If you qualify for participation, you will have blood work done to measure your cholesterol and other fat levels through a lipid panel. You will be provided with these results free of charge at the conclusion of the study.

Phase 2

You will receive the study medication. Half of the participants will receive the actual product we are investigating and half will receive a placebo (inactive/dummy pill). Neither you nor the investigators will not know which one you are given until the end of the study. During the 4th and 12th weeks, you will be asked to keep a diary (similar to the first one) of your hot flashes.

Phase 3

At the end of the 12 week study period, you will return to the study center. The second blood draw will be done to monitor any changes. This will conclude your participation. You will be sent a copy of your cholesterol profiles and FSH levels approximately 2 weeks after you complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal females (no periods for over 6 months)
* Documented Serum FSH level>20
* Positive urine FSH test
* Hot flashes, on average five a day
* A 2 week pre study washout period of exclusion criteria

Exclusion Criteria:

* No EPT/ET
* OTC supplements: ex; soy, black cohosh, flax, bellergal, primrose oil, vitamin E, red clover
* Excessive smoking > 1ppd
* Anti seizure medications
* Clonidine
* Effexor
* More than 2 servings of fish per week

Max Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The decrease in the severity in hot flashes. | 3 months

SECONDARY OUTCOMES:
Improvement in lipid profile | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Parastoo Farhady, MD, Principal Investigator — Chrisitiana care Health Systems
Locations (1):
- Christiana Care Health Systems, Newark, Delaware, United States